CLINICAL TRIAL: NCT01112059
Title: A Randomized Trial of Doxycycline to Reduce Sputum MMP-9 Activity in Adult CF Patients Hospitalized for Pulmonary Exacerbations
Brief Title: Trial of Doxycycline to Reduce Sputum MMP-9 Activity in Adult Cystic Fibrosis (CF) Patients
Acronym: DOXY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Amit Gaggar, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F081024004
Record Dates: First submitted 2010-04-20; First posted 2010-04-28 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients given placebo twice a day for 8 days at beginning of inpatient CF exacerbation
  Interventions: Other: placebo
- doxycycline (Active Comparator): Patients given doxycycline 100 mg tablet twice a day for 8 days at the beginning of inpatient CF exacerbation
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — 100 mg twice a day for 8 days
  Arms: doxycycline
Other: placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the role of a well-known and well-tolerated antibiotic, doxycycline, in the treatment of cystic fibrosis patients who are hospitalized. This antibiotic does not effectively treat the bacteria in airways of cystic fibrosis patients, but may reduce the activity of inflammatory molecules in the disease.

DETAILED DESCRIPTION:
One molecule that is inhibited by doxycycline is matrix metalloprotease-9, which is emerging as an important mediator of lung inflammation and damage in cystic fibrosis. We hypothesize that the addition of treatment with doxycycline in CF inpatients will reduce MMP-9 activity and inflammatory markers in the sputum of cystic fibrosis patients compared to CF patients not treated with doxycycline.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis
* Hospitalization for Pulmonary exacerbation

Exclusion Criteria:

* Significant GI illness
* Participation in another Investigational Protocol
* Allergies to Doxycycline
* Sputum Culture only positive for Staphylococcus aureus,
* Pregnant or Nursing
* Unwilling to use effective birth control
* Elevated LFT's greater than 3x the upper limit of normal
* Creatinine greater than 1.5x the upper limit of normal
* Lung transplantation
* Substance abuse within 30 days of screening

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Gaggar, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu X, Abdalla T, Bratcher PE, Jackson PL, Sabbatini G, Wells JM, Lou XY, Quinn R, Blalock JE, Clancy JP, Gaggar A. Doxycycline improves clinical outcomes during cystic fibrosis exacerbations. Eur Respir J. 2017 Apr 5;49(4):1601102. doi: 10.1183/13993003.01102-2016. Print 2017 Apr. PMID 28381428

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Doxycycline
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Doxycycline | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (9.4) | 29.1 (8.9) | 28.2 (9.1)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 13 | 12 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Examines tolerability and safety with focus on adverse events (AEs) and serious adverse events (SAEs)
Time Frame: 1 month from enrollment
Measure: Number; unit: adverse events
Groups:
- Placebo: placebo: placebo
  No SAEs noted in this group, 4 total AEs recorded.
Arm/Group | Placebo | Doxycycline
Number analyzed (Participants) | 19 | 20
adverse events | 5 | 5

2. Primary Outcome: Matrix Metalloprotease-9 (MMP-9) Protein Levels in Sputum
Description: Mean sputum matrix metalloprotease-9 (MMP-9) levels measured at the end of therapy
Time Frame: 8 days past baseline
Measure: Mean (Standard Deviation); unit: ng/mg total protein
Groups:
- Placebo: placebo for 8 days
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 20 | 19
ng/mg total protein | 4034 (3459) | 8837 (14752)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 0.5, 95% CI 2-sided [0.128 to 0.633]

3. Secondary Outcome: Mean Sputum Matrix Metalloprotease-9 (MMP-9) Activity End of Treatment
Description: Measurement of endogenous active matrix metalloprotease-9 (MMP-9) in the sputum
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: ng/mg total protein
Arm/Group | Placebo | Doxycycline
Number analyzed (Participants) | 19 | 20
ng/mg total protein | 12683 (35275) | 3224 (2683)

4. Secondary Outcome: Mean Change in Pulmonary Function Over Treatment Duration
Description: Observe change in FEV1% predicted from beginning to end of study
Time Frame: Baseline to end of inpatient clinical exacerbation (average 14 days)
Measure: Mean (Standard Deviation); unit: Percentage of predicted FEV1
Arm/Group | Placebo | Doxycycline
Number analyzed (Participants) | 19 | 20
Percentage of predicted FEV1 | 6.9 (10.4) | 10.0 (6.8)

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | Placebo | Doxycycline
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 5/19 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Doxycycline (N=20)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Increased cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
tingling of lips (General disorders) | 0 (0) | 1 (1) — Self-limited tingling of lips
Headache (General disorders) | 0 (0) | 1 (1)
Pelvic pain (Renal and urinary disorders) | 1 (1) | 0 (0) — Transient pelvic pain
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Although the study has a relatively large number of subjects, this was a single center trial. In addition, it is possible that the protein readouts are mediated by modulating the dysregulated protease activity in the airway.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No